CLINICAL TRIAL: NCT03936062
Title: Replication of the TECOS Diabetes Trial in Healthcare Claims
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-TECOS
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate; Sulfonylurea Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2nd Generation SUs: Reference group
  Interventions: Drug: Sulfonylurea
- Sitagliptin: Exposure group
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin dispensing claim is used as the exposure
  Groups: Sitagliptin
Drug: Sulfonylurea — 2nd generation sulfonylurea dispensing claim is used as the reference
  Groups: 2nd Generation SUs

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Inclusion Criteria:

* Patients with a diagnosis of T2DM (ICD-9 Dx code of 250.x0 or 250.x2; ICD-10 Dx code of E11.x) in the 6 months prior to drug initiation
* Metformin, pioglitazone, or a sulfonylurea (monotherapy or any dual combination) for each day in the prior 3 months
* Any insulin use for each day in the prior 3 months
* 2 outpatient visits
* Patient is ≥50 years of age
* History of a major clinical manifestation of coronary artery disease (i.e., MI, surgical or percutaneous [balloon and/or stent] coronary revascularization procedure
* Ischemic cerebrovascular disease, including:

  * History of ischemic stroke. Strokes not known to be hemorrhagic will be allowed as part of this criterion;
  * Occlusion and stenosis of carotid artery without mention of cerebral infarction as History of carotid arterial disease as documented by ≥50% stenosis documented by carotid ultrasound, magnetic resonance imaging (MRI), or angiography, with or without symptoms of neurologic deficit
  * Peripheral arterial stenting or surgical revascularization, Lower extremity amputation, and Ankle brachial pressue index <0.9 as: Atherosclerotic peripheral arterial disease, as documented by objective evidence such as amputation due to vascular disease, current symptoms of intermittent claudication confirmed by an anklebrachial pressure index or toe brachial pressure index less than 0.9, or history of surgical or percutaneous revascularization procedure.
* Encounter for contraceptive management and oral contraceptives as Female patients agree to use an effective method of contraception or must not otherwise be at risk of becoming pregnant.

Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or a history of ketoacidosis.
* Patient has a history of ≥2 episodes of severe hypoglycemia during the 12 months prior to enrollment. Severe hypoglycemia (hypoglycemia requiring assistance) refers to instances in which the patient was sufficiently disoriented or incapacitated as to require help from another individual or from medical personnel (whether or not this assistance was actually provided).
* Patient has taken an approved or investigational DPP-4 inhibitor agent (eg, sitagliptin, alogliptin, saxagliptin, or vildagliptin), GLP-1 analogues (eg, exenatide, exenatide LAR, or liraglutide), or a thiazolidinedione other than pioglitazone within the past 3 months.
* Patient has cirrhosis of the liver, as assessed by medical history.
* Pregnancy or planned pregnancy during the trial period.
* Exclude patients with a combined comorbidity score >95th percentile as Patient has medical history that indicates a life expectancy of b2 years or might limit the individual's ability to take trial treatments for the duration of the study.

Ages: 50 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing sitagliptin to the 2nd generation sulfonylurea antidiabetic class as a proxy for placebo, since this class of antidiabetic drugs is not known to have an impact on the outcome of interest. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of sitagliptin or a comparator drug (index date). Follow-up for the outcome (4P-MACE), begins the day after drug initiation. As in the trial, patients are allowed to take other antidiabetic medications during the study. Eligible cohort entry dates: 10/17/2006-12/31/2016 (market availability of sitagliptin in the U.S. started on 10/17/2006). For Optum, 10/17/2006-9/30/201.
Sampling Method: Non-Probability Sample
Enrollment: 349476 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Relative hazard of composite outcome of ACS/unstable angina, Stroke, MI, and Mortality | Through study completion (a median of 118 days)
  Relative hazard of composite outcome of ACS/unstable angina, MI, stroke, and mortality - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Womens
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Franklin JM, Patorno E, Desai RJ, Glynn RJ, Martin D, Quinto K, Pawar A, Bessette LG, Lee H, Garry EM, Gautam N, Schneeweiss S. Emulating Randomized Clinical Trials With Nonrandomized Real-World Evidence Studies: First Results From the RCT DUPLICATE Initiative. Circulation. 2021 Mar 9;143(10):1002-1013. doi: 10.1161/CIRCULATIONAHA.120.051718. Epub 2020 Dec 17. PMID 33327727

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT03936062/Prot_SAP_001.pdf